CLINICAL TRIAL: NCT02695628
Title: Assessment of Treatment-Induced Tissue Hypoxia After Transcatheter Arterial Embolization of Hepatocellular Carcinoma: A Feasibility Study With [18F]FMISO PET/CT
Brief Title: [18F]FMISO PET/CT After Transcatheter Arterial Embolization in Imaging Tumors in Patients With Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-29768; NCI-2016-00041 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEP0055 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2016-02-24; First posted 2016-03-01 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Adult Liver Carcinoma; Liver Cirrhosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis | interventions — fluoromisonidazole; Tomography, X-Ray Computed; Tomography; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (18F-fluoromisonidazole, PET/CT, embolization) (Experimental): Patients undergo transcatheter arterial embolization. Patients also receive 18F-fluoromisonidazole IV and undergo PET/CT scans 4 weeks prior to embolization treatment and in the 20 hours following completion of treatment.
  Interventions: Drug: 18F-Fluoromisonidazole; Procedure: Arterial Embolization; Diagnostic Test: Computed Tomography; Diagnostic Test: Positron Emission Tomography

INTERVENTIONS:
Drug: 18F-Fluoromisonidazole — Undergo [18F] FMISO PET/CT
  Other Names: 18F-MISO; 18F-Misonidazole; FMISO
Procedure: Arterial Embolization — Undergo transcatheter arterial embolization
  Other Names: TAE; Transarterial Embolization
Diagnostic Test: Computed Tomography — Undergo [18F] FMISO PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Diagnostic Test: Positron Emission Tomography — Undergo [18F] FMISO PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial studies how well 18F-fluoromisonidazole ([18F]FMISO) positron emission tomography (PET)/computed tomography (CT) works after transcatheter arterial embolization in imaging tumors in patients with liver cancer. Transcatheter arterial embolization blocks blood flow to tumor cells by inserting tiny foreign particles into an artery near the tumor. [18F]FMISO is a type of radioimaging agent that binds to large molecules in tumor cells that have a low level of oxygen, and the radiation given off by [18F]FMISO is picked up by a PET scan and this may help researchers learn whether changes occur in the tumors after treatment, which can help decide how well the treatment worked earlier than is currently possible

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the variability of 18F FMISO uptake in hepatocellular carcinoma (HCC) tumors compared to normal liver after transcatheter arterial embolization by determining the difference in the mean of the maximum standardized uptake value (SUVmax) and tumor-to-liver ratio (TLR) of a region of normal liver and of up to 5 index tumors.

SECONDARY OBJECTIVES:

I. Determine if areas of tumor recurrence as determined by CT or magnetic resonance imaging (MRI) within a 6 month period after transcatheter arterial embolization show evidence of increased 18F FMISO labeling on the initial post treatment 18F FMISO PET/CT.

II. Determine the variability in SUVmax and TLR of untreated (non embolized) HCC lesions compared to normal liver by determining the difference in the mean of the SUVmax and TLR of normal liver and tumor.

III. Determine any toxicities related to [18F]FMISO use for PET/CT.

OUTLINE:

Patients undergo transcatheter arterial embolization. Patients also receive 18F-fluoromisonidazole intravenously (IV) and undergo PET/CT scans within 4 weeks prior to embolization treatment and in the 20 hours following completion of treatment.

After completion of treatment, patients are followed up at 2 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Histopathologic or imaging and clinical features of tumor(s) diagnostic for hepatocellular carcinoma with at least one tumor >= 1.5 cm; imaging features diagnostic for hepatocellular carcinoma will be defined as Liver Imaging Reporting and Data System (LIRADS) 4 or greater
* Total bilirubin < 3.0
* Child Pugh A or B
* Tumor amenable to transcatheter arterial embolization
* Able to provide informed consent

Exclusion Criteria:

* Uncontrolled large ascites
* Main or segmental portal vein thrombosis
* Locoregional treatment of hepatocellular carcinoma within the prior 3 months or chemotherapy within the previous 3 months
* Inability or contraindication to undergo transcatheter arterial embolization
* Inability to lay flat for at least 2 consecutive hours
* Severe acute illness
* Uncontrolled chronic illness such as hypertension, diabetes, or heart failure
* Contraindication to CT or MRI contrast
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Shah, Principal Investigator — Stanford Cancer Institute
Locations (1):
- VA Palo Alto Healthcare System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah RP, Laeseke PF, Shin LK, Chin FT, Kothary N, Segall GM. Limitations of Fluorine 18 Fluoromisonidazole in Assessing Treatment-induced Tissue Hypoxia after Transcatheter Arterial Embolization of Hepatocellular Carcinoma: A Prospective Pilot Study. Radiol Imaging Cancer. 2022 May;4(3):e210094. doi: 10.1148/rycan.210094. PMID 35485937

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (18F-fluoromisonidazole, PET/CT, Embolization)
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (18F-fluoromisonidazole, PET/CT, Embolization)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (5.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Maximum Standardized Uptake Value (SUVmax) in Tumor vs Normal Tissue [Mean (Standard Deviation); unit: Ratio] — Before participants undergo transcatheter arterial embolization (TACE), ie, at baseline, 18F-fluoromisonidazole (18F-FMISO) positron emission tomography (PET)/computed tomography (CT) scans were conducted. Maximum standardized uptake value (SUVmax) were determined at the tumor lesion and in normal tissue, represented by liver. The variability of 18F-FMISO uptake in hepatocellular carcinoma (HCC) tumors before treatment was assessed as the ratio of the SUVmax as observed in the tumor vs liver (tumor-to-liver ratio, TLR). The data is reported as the mean TLR, with standard deviation.
  Ratio | 0.71 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: Post-treatment Maximum Standardized Uptake Value (SUVmax) in Tumor and Normal Tissue
Description: All participants undergo transcatheter arterial embolization (TACE) and 18F-fluoromisonidazole (18F-FMISO) positron emission tomography (PET)/computed tomography (CT) scans were conducted. Maximum standardized uptake value (SUVmax) were determined at the tumor lesion and in normal tissue, represented by liver. The variability of 18F-FMISO uptake in hepatocellular carcinoma (HCC) tumors post-TACE was assessed as the ratio of the SUVmax as observed in the tumor vs liver (tumor-to-liver ratio, TLR). The outcome is reported as the mean TLR, with standard deviation.
Time Frame: 24 hours
Population: Due to withdrawal, not all participants completed for this outcome.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Diagnostic (18F-fluoromisonidazole, PET/CT, Embolization)
Number analyzed (Participants) | 4
Ratio | 0.76 (0.14)

2. Secondary Outcome: Maximum Standardized Uptake Value (SUVmax) at Lesion Sites With and Without Tumor Recurrence
Description: Follow-up 18F-fluoromisonidazole (18F-FMISO) positron emission tomography (PET)/computed tomography (CT) scans were to be conducted within 6 months or at the time of tumor recurrence. Maximum standardized uptake value (SUVmax) were determined at the tumor lesion and in normal tissue, represented by liver. The variability of 18F-FMISO uptake at the hepatocellular carcinoma (HCC) tumor lesion site post-TACE was assessed as the mean difference in the ratio of the SUVmax as observed in the tumor vs liver (tumor-to-liver ratio, TLR), between lesions that recurred, and those that did not. The outcome is reported as the mean TLR, with standard deviation.
Time Frame: Up to 6 months
Population: Follow-up 18F-fluoromisonidazole (18F-FMISO) positron emission tomography (PET) scans at the time of tumor recurrence were not conducted.
Arm/Group | Diagnostic (18F-fluoromisonidazole, PET/CT, Embolization)
Number analyzed (Participants) | 0

3. Secondary Outcome: Adverse Events Related to 18F-fluoromisonidazole (18F-FMISO)
Description: Toxicity to 18F-fluoromisonidazole (18F-FMISO) was assessed by the number of adverse events that occurred within 18 hours of administration (about 10 half-lives), that were also unanticipated and related to 18F-FMISO. The outcome is reported as the number of adverse events that were unanticipated and related to 18F-FMISO, a number without dispersion.
Time Frame: 18 hours
Population: All participants are included for this outcome.
Measure: Number; unit: Number of adverse events
Arm/Group | Diagnostic (18F-fluoromisonidazole, PET/CT, Embolization)
Number analyzed (Participants) | 5
Number of adverse events | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Diagnostic (18F-fluoromisonidazole, PET/CT, Embolization)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (18F-fluoromisonidazole, PET/CT, Embolization) (N=5)
Fatigue (General disorders) | 4 (4)
Hepatic pain (Hepatobiliary disorders) | 2 (3)
Edema limbs (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Infections and infestations -Other, Cellulitis (Infections and infestations) | 1 (1)
Hepatobiliary disorders -Other, increased liver functions (Hepatobiliary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT02695628/Prot_SAP_000.pdf